CLINICAL TRIAL: NCT00840840
Title: An Open-Label, Single-Dose, Two-Way Crossover Bioequivalence Study of Two Oral Suspension Formulations of Amoxicillin/Clavulanate Potassium, 600/42.9 mg/5 mL in Healthy Subjects, Under Fed Conditions
Brief Title: 600 mg Amoxicillin/42.9 mg Clavulanate Postassium /5 mL Suspension Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 02-544
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 600 mg Amoxicillin/42.9 mg Clavulanate Postassium /5 mL
- 2 (Active Comparator)
  Interventions: Drug: Augmentin ES-600™

INTERVENTIONS:
Drug: 600 mg Amoxicillin/42.9 mg Clavulanate Postassium /5 mL — 1 x 600 mg/42.9 mg/5 mL, single-dose fasting
  Arms: 1
Drug: Augmentin ES-600™ — 1 x 600 mg/42.9 mg/5 mL, single-dose fasting
  Arms: 2

SUMMARY:
The purpose of this study is to assess the bioequivalence between Amoxicillin/Clavulanate Potassium Oral Suspension 600/42.9 mg/5 mL and Augmentin ES-600 Oral Suspension, 600/42.9 mg/5 mL in healthy, male and female subjects, under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male or non-pregnant, non-lactating female subjects, 18 years of age and over.
* Body weight within ±15% of the appropriate weight range published in 1993 by Metropolitan Life Insurance Company, Statistical Bureau and body-mass index (BMI) less than 30.
* Negative for:

  * HIV
  * Hepatitis B and C
  * Urine drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).
  * Cotinine (urine test)
  * Breath alcohol (Breathalyzer)
  * HCG (females only)
* No significant diseases or clinically significant abnormal laboratory values.
* No clinically significant findings in the physical examination.
* No clinically significant findings in vital sign measurements and 12-lead electrocardiogram (ECG).
* Informed of the nature of the study and give written consent prior to receiving any study medication.
* Female subjects: surgically steril, post-menopausal or practicing a recognized safe method of contraception (abstention, oral or implanted contraceptives, intra-uterine device or consistent condom plus spermicide use).

Exclusion Criteria:

* Known history or presence of any disease or condition which might compromise the following body systems: immunologic, endocrine, renal, cardiovascular, respiratory, hematologic, gastrointestinal, neurologic, hepatic, psychiatric or dermatologic
* More specifically: history or presence of significant: sensitivity to multiple allergens, diarrhea, stomach or intestinal disease, mononucleosis, renal or hepatic dysfunction and asthma.
* Known or suspected carcinoma.
* Known history or presence of:

  * Hypersensitivity or idiosyncratic reaction to amoxicillin, clavulanic acid, penicillin, cephalosporins and/or any other β-lactamase inhibitors.
  * Clavulin-associated jaundice/hepatic dysfunction.
  * Alcoholism within last 12 months.
  * Drug dependence and/or substance abuse.
  * Use of tobacco or nicotine-containing products, within last 12 months.
* On a special diet within 4 weeks prior to drug administration (i.e. a deliberate change in diet for any reason).
* Participation in another clinical trial or received an investigational product in the previous 30 days prior to drug administration.
* Donation up to 250 mK of blood in the previous 30 days, 251-500 mKL in the previous 45 days, 501-750 mL in the previous 60 days or above 750 mL in the previous 90 days prior to study start.
* Requirement of any medication, (prescription and/or over-the-counter) or dietary supplements on a routine basis, with the exception of occasional use of acetaminophen and oral or implanted contraceptives.
* Difficulty fasting or consuming the standard prescribed meals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Ph.D., Principal Investigator — Pharma Medica Research
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Test First: Amoxicillin and Clavulante Potassium for Oral Suspension, 600/42.9 mg/5mL test product dosed in first period followed by AugmentinES-600™ for Oral Suspension 600/42.9 mg/5mL reference product dosed in second period
- Reference First: AugmentinES-600™ for Oral Suspension 600/42.9 mg/5mL reference product dosed in first period followed by Amoxicillin and Clavulante Potassium for Oral Suspension 600/42.9 mg/5mL test product dosed in second period
Period: Period 1
Arm/Group | Test First | Reference First
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test First | Reference First
Started | 23 (One subject was withdrawn due to AE after Period 1) | 24
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test First | Reference First | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 20 | 18 | 38
  Black | 3 | 4 | 7
  Asian | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based on Cmax for Amoxicillin
Description: Cmax - Maximum Observed Concentration
Time Frame: Blood samples collected over 14 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Amoxicillin Clavulanate: Amoxicillin and Clavulante Potassium for Oral Suspension, 600/42.9 mg/5mL test product dosed in either period
- AugmentinES-600™: AugmentinES-600™ for Oral Suspension 600/42.9 mg/5mL reference product dosed in either period
Arm/Group | Amoxicillin Clavulanate | AugmentinES-600™
Number analyzed (Participants) | 47 | 47
ng/mL | 7331.46 (1414.94) | 7235.76 (1434.42)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanate vs AugmentinES-600™; Test type: Non-Inferiority or Equivalence — ANOVA; Test/Reference Ratio of the mean x 100 = 101.45, 90% CI [97.71 to 105.33] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: Bioequivalence Based on AUC0-inf for Amoxicillin
Description: AUC0-inf - Area under the concentration-time curve from time zero to infinity (extrapolated)
Time Frame: Blood samples collected over 14 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanate | AugmentinES-600™
Number analyzed (Participants) | 47 | 47
ng*h/mL | 27318.54 (4774.49) | 26515.59 (4691.18)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanate vs AugmentinES-600™; Test type: Non-Inferiority or Equivalence — ANOVA; Test/Reference Ratio of the mean x 100 = 103.05, 90% CI [101.25 to 104.88] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: Bioequivalence Based on AUC0-t for Amoxicillin
Description: AUC0-t - Area under the concentration-time curve from time zero to time of last non-zero concentration
Time Frame: Blood samples collected over 14 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanate | AugmentinES-600™
Number analyzed (Participants) | 47 | 47
ng*h/mL | 26662.17 (4754.01) | 25906.24 (4662.03)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanate vs AugmentinES-600™; Test type: Non-Inferiority or Equivalence — ANOVA; Test/Reference Ratio of the mean x 100 = 102.94, 90% CI [101.08 to 104.83] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

4. Primary Outcome: Bioequivalence Based on Cmax for Clavulanic Acid
Description: Cmax - Maximum Observed Concentration
Time Frame: Blood samples collected over 14 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amoxicillin Clavulanate | AugmentinES-600™
Number analyzed (Participants) | 47 | 47
ng/mL | 516.42 (197.44) | 507.38 (162.09)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanate vs AugmentinES-600™; Test type: Non-Inferiority or Equivalence — ANOVA; Test/Reference Ratio of the mean x 100 = 99.68, 90% CI [92.41 to 107.52] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

5. Primary Outcome: Bioequivalence Based on AUC0-inf for Clavulanic Acid
Description: AUC0-inf - Area under the concentration-time curve from zero to infinity (extrapolated)
Time Frame: Blood samples collected over 14 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanate | AugmentinES-600™
Number analyzed (Participants) | 47 | 47
ng*h/mL | 1335.73 (628.13) | 1283.73 (508.17)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanate vs AugmentinES-600™; Test type: Non-Inferiority or Equivalence — ANOVA; Test/Reference Ratio of the mean x 100 = 101.48, 90% CI [94.73 to 108.71] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

6. Primary Outcome: Bioequivalence Based on AUC0-t for Clavulanic Acid
Description: AUC0-t - Area under the concentration-time curve from time zero to time of last non-zero concentration
Time Frame: Blood samples collected over 14 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/h/mL
Arm/Group | Amoxicillin Clavulanate | AugmentinES-600™
Number analyzed (Participants) | 47 | 47
ng/h/mL | 1241.09 (627.50) | 1195.82 (503.91)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanate vs AugmentinES-600™; Test type: Non-Inferiority or Equivalence — ANOVA; Test/Reference Ratio of the mean x 100 = 100.17, 90% CI [91.95 to 109.13] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is not permitted to discuss or publish trial results.